CLINICAL TRIAL: NCT01179243
Title: Observation of the Prevalence of Sublingual Microcirculatory Alterations With SDF Imaging in Intensive Care Patients
Brief Title: Prevalence of Microcirculatory Alterations in Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, E.C. Boerma, MD PhD, Frisius Medisch Centrum
Other Study IDs: TPO 702
Record Dates: First submitted 2010-08-03; First posted 2010-08-11 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Critical Illness
Keywords: microcirculatory alterations; SDF imaging
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intensive care patients: no interventions

SUMMARY:
Recent research has focused on the investigation of sublingual microcirculatory alterations in different patient categories, like cardiac surgery and sepsis. The microcirculation plays a pivotal role in tissue oxygenation and can be non invasively visualized by sidestream dark field (SDF) imaging.

The objective is to carry out a international multi center study to investigate the prevalence of microcirculatory alterations in intensive care patients. Up to the present time, a comprehensive prevalence study like this has not been carried out.

DETAILED DESCRIPTION:
Visualization of the sublingual microcirculation at a fixed time point with SDF- or OPS-imaging in all adult patients of participating intensive care units, regardless of their underlying disease. Concurrently, data on both patient characteristics (e.g. severity of illness, treatment) and ICU characteristics will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* > 18
* informed consent

Exclusion Criteria:

* injury to the maxillofacial area
* recent maxillofacial injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
microcirculatory alterations related to underlying illness, expressed as - amongst others- microvascular flow index (MFI), proportion of perfused vessels (PPV). | 24 hours

SECONDARY OUTCOMES:
microcirculatory alterations related to: hospital/intensive care length of stay mortality severity of illness | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: E.C. Boerma, MD, PhD, Principal Investigator — Medical Centre Leeuwarden, the Netherlands
Locations (4):
- Netherlands (4):
  - OLVG, Amsterdam
  - Gelre Ziekenhuis Apeldoorn, Apeldoorn
  - Medical Centre Leeuwarden, Leeuwarden
  - Erasmus MC Rotterdam, Rotterdam

REFERENCES:
- [Derived] Vellinga NAR, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, van der Voort PHJ, Dondorp AM, Bafi T, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Bakker J, Ince C; microSOAP study group. Mildly elevated lactate levels are associated with microcirculatory flow abnormalities and increased mortality: a microSOAP post hoc analysis. Crit Care. 2017 Oct 18;21(1):255. doi: 10.1186/s13054-017-1842-7. PMID 29047411
- [Derived] Vellinga NA, Boerma EC, Koopmans M, Donati A, Dubin A, Shapiro NI, Pearse RM, Machado FR, Fries M, Akarsu-Ayazoglu T, Pranskunas A, Hollenberg S, Balestra G, van Iterson M, van der Voort PH, Sadaka F, Minto G, Aypar U, Hurtado FJ, Martinelli G, Payen D, van Haren F, Holley A, Pattnaik R, Gomez H, Mehta RL, Rodriguez AH, Ruiz C, Canales HS, Duranteau J, Spronk PE, Jhanji S, Hubble S, Chierego M, Jung C, Martin D, Sorbara C, Tijssen JG, Bakker J, Ince C; microSOAP Study Group. International study on microcirculatory shock occurrence in acutely ill patients. Crit Care Med. 2015 Jan;43(1):48-56. doi: 10.1097/CCM.0000000000000553. PMID 25126880